CLINICAL TRIAL: NCT00715429
Title: Nocturnal Leg Cramps in the Elderly: Randomized Controlled Trial of Ergocalciferol (Vitamin D2) for a Painful and Distressing Problem
Brief Title: Vitamin D for Painful Nocturnal Leg Cramps
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We exhausted potential candidates before reaching goal of 70; recruited 29, 13 completed the study
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2007-0255
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Leg Cramps, Nocturnal
Keywords: Leg cramps; vitamin D deficiency
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Vitamin D Deficiency | interventions — Vitamin D; Ergocalciferols; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vitamin D 50,000 U/d x 10d, + vitamin D 50,000 U weekly 7 wks (Experimental): Vitamin D arm
  Interventions: Drug: vitamin d
- placebo x 10d, + placebo weekly 7 wks (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vitamin d — After a two-week wash-in, subjects will take a vitamin D capsule (50,000 units) once daily for 10 days, followed by a once weekly vitamin D (50,000 units) maintenance dose for 7 weeks.
  Other Names: ergocalciferol
  Arms: vitamin D 50,000 U/d x 10d, + vitamin D 50,000 U weekly 7 wks
Drug: placebo — After a two-week wash-in, subjects will take a placebo capsule once daily for 10 days, followed by a once weekly maintenance dose for 7 weeks.
  Other Names: lactose
  Arms: placebo x 10d, + placebo weekly 7 wks

SUMMARY:
1. Research question: Does vitamin D reduce the frequency and severity of nocturnal leg cramps in older persons who previously took quinine for leg cramps?
2. Experimental Design: This is a randomized, double blind, placebo controlled study of 70 men and women veterans receiving care at the Madison VA Medical Center(VAMC) or at the University of Wisconsin Hospitals and Clinics (UWHC). Individuals age 50 or more who have previously taken quinine for nocturnal leg cramps and meeting baseline criteria are eligible to enroll. Enrollees meeting laboratory criteria, including low-normal vitamin D levels, will undergo a 2-week "diary run-in" period to confirm cramp frequency. Those who report two or more leg cramps in each week will continue in the study and will be randomized to vitamin D or placebo. After a two-week wash-in, subjects will take a vitamin D capsule (50,000 units) once daily for 10 days, followed by a once weekly vitamin D (50,000 units) maintenance dose for 7 weeks. Subjects will record by diary the number and severity of leg cramps from the start of the "diary run-in" until a week after the last dose of study drug. Study investigators will call subjects at scheduled intervals to assess compliance, tolerability, and diary use.
3. Major risks to subjects: No major risks are anticipated. Excessive vitamin D can increase blood calcium levels (hypercalcemia), with symptoms such as thirst, nausea, and weakness. However, symptomatic hypercalcemia has not been reported except for those taking more than 40,000 units daily for several months. This is far above the cumulative dose in our study.
4. Potential benefits: Subjects may not receive any benefit. Vitamin D may alleviate leg cramps for subjects who receive it.
5. Consent Procedure: Flyers describing the study and telephone contact information will be mailed to patients who have received quinine during the period 2002-2007. The PI or Co-PI will return calls to describe the study and answer any questions. For persons meeting preliminary (pre-lab) study criteria, two copies of the consent form will be mailed, with the patient mailing back one signed consent to the PI.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial to determine if oral vitamin D administration reduces the number or severity of nocturnal leg cramps, compared to placebo. Symptom diaries will be used throughout the study to assess frequency and severity of cramps. We will enroll a total of 70 men and women at least 50 years of age who have nocturnal leg cramps at least twice weekly and have previously received quinine for this. Those meeting baseline laboratory criteria and who report at least two leg cramps per week in a two-week "diary run-in" period will be randomized to vitamin D or placebo. Baseline, mid-study, and final laboratory testing will assess any changes in 25-hydroxyvitamin D(OHD) and related variables (25-hydroxyvitamin D is the best measure of vitamin D status.) The time from the beginning of the diary run-in through the final dose of drug and last labs,will be about 14 weeks.

Optimal vitamin D status for health is unknown, although many experts aim for serum 25-hydroxyvitamin D of 35-40 ng/ml. Subjects in this study randomized to vitamin D will take a vitamin D capsule (50,000 units) once daily for 10 days, followed by a once weekly vitamin D (50,000 units) maintenance dose for 7 weeks. Based on published literature on the ability of vitamin D to raise serum 25-OHD over time, we estimate that the loading doses will "boost" levels after 10 days by an increment of ~40ng/ml (up to ~65 ng/mL total, starting with a typical person's baseline of 25ng/ml). This achieved level of 65 is within the reference range of our VA's reference range of 20-100. (In the PI's experience, most veterans without special D supplementation have baseline levels between 15 and 40).

ELIGIBILITY:
Inclusion Criteria:

* One or more prescription for quinine at the Madison VA in the last 5 years, or else be a UWHC (U Wisconsin Health Clinics) patient whose UWHC medication list had quinine listed in the last five years
* At least 50 years of age, with women being past menopause. This is defined as the woman reporting no periods in the last 12 consecutive months or longer.
* Leg cramps listed in medical record,
* Ability & willingness to give informed consent,
* Stable estimated Glomerular filtration rate (GFR)>35 ml/min for the prior 6 mos,
* No change in diuretic therapy in last 3 months,
* Stable pattern of two or more cramps per week for past three months,
* Ability to complete daily diary entry,
* Post-consent: serum 25-OH of 20-45 ng/mL, albumin- corrected calcium <10.3 mg/dL, and urine calcium/creatinine ratio <0.25.

Exclusion Criteria:

* Not receiving primary care at Madison VAMC, or at UWHC
* Hyperparathyroidism (1°, 2°, or 3°),
* Osteomalacia ,
* Paget's disease,
* Metastatic cancer,
* Taking vitamin D 50,000 units capsules,
* Serum Ca++ >10.3 mg/dL in subject chart,
* Sarcoidosis or tuberculosis, and
* Peripheral vascular disease or other condition confounding assessment of cramps.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Elliott, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants got excluded from the study due to not fulfilling the inclusion criteria.
Period: Overall Study
Arm/Group | Vitamin D 50,000 U/d x 10d, + Vitamin D 50,000 U Weekly 7 Wks | Placebo x 10d, + Placebo Weekly 7 Wks
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Did not complete the study diary | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D 50,000 U/d x 10d, + Vitamin D 50,000 U Weekly 7 Wks | Placebo x 10d, + Placebo Weekly 7 Wks | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Full Range); unit: years] | 78 [64 to 87] | 73 [62 to 79] | 76 [62 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
Leg cramp frequency mean over 2 week prestudy [Mean (Standard Deviation); unit: cramps/day] — Eligibility requirements included having at least two cramps weekly.
  cramps/day | 0.74 (0.56) | 1.27 (1.15) | 1.005 (0.855)
25-hydroxyvitamin D concentration [Mean (Standard Deviation); unit: ng/ml] — Eligibility requirements included having 25-hydroxyvitamin D concentration between 20 and 45 ng/ml.
  ng/ml | 38 (6) | 34 (8) | 37 (7)
Serum calcium [Mean (Standard Deviation); unit: mg/dL] — Eligibility requirements included having normal serum calcium ranging from 8.5-10.2 mg/dL.
  mg/dL | 9.0 (0.2) | 9.1 (0.4) | 9.05 (0.3)
Urine calcium /creatinine ratio [Mean (Standard Deviation); unit: ratio] | 0.09 (0.10) | 0.10 (0.08) | .095 (.09)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min] | 69 (19.6) | 81 (25) | 75 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Nocturnal Leg Cramp Rate
Description: Difference in number of leg cramps per day during treatment period compared to baseline period.
  Participants will undergo a 2-week "diary run-in" period to confirm cramp frequency. After a 2 week wash-in, subjects will take a vitamin D capsule (50,000 units) once daily for 10 days, followed by a once weekly vitamin D (50,000 units) maintenance dose for 7 weeks. Subjects will record by diary the number and severity of leg cramps from the start of the "diary run-in" until 1 week after the last dose of study drug/placebo.
Time Frame: baseline and 77 day
Measure: Mean (Standard Deviation); unit: cramps/day
Groups:
- Vitamin D: Vitamin D
  vitamin d: After a two-week wash-in, subjects will take a vitamin D capsule (50,000 units) once daily for 10 days, followed by a once weekly vitamin D (50,000 units) maintenance dose for 7 weeks.
- Placebo: Placebo
  placebo: After a two-week wash-in, subjects will take a placebo capsule once daily for 10 days, followed by a once weekly maintenance dose for 7 weeks.
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 6
cramps/day | 0.07 (0.28) | -0.05 (0.35)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.27, t-test, 2 sided — Daily cramp rate at baseline& on treatment, were calculated as % of each subjects total # of cramps, for comparison among subjects. Change in % cramp rates from baseline to treatment was computed for each subject in vit D and placebo groups; T test was used to compare the change in % cramp rate from baseline to treatment for each subject in each treatment group

2. Secondary Outcome: Serum Calcium Level
Description: Serum calcium was measured to detect any possible correlation between high dose of Vitamin D and hypercalcemia. Hypercalcemia is defined as a serum calcium level greater than 10.5 mg/dL.
Time Frame: Day 77
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 7 | 6
mg/dL | 9.4 (0.3) | 9.2 (0.4)

ADVERSE EVENTS:
Arm/Group | Vitamin D 50,000 U/d x 10d, + Vitamin D 50,000 U Weekly 7 Wks | Placebo x 10d, + Placebo Weekly 7 Wks
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 3/7 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D 50,000 U/d x 10d, + Vitamin D 50,000 U Weekly 7 Wks (N=7) | Placebo x 10d, + Placebo Weekly 7 Wks (N=6)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — diabetic patient took too much insulin, dose was lowered
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — long term undiagnosed anemia, sees hematology clinic
post traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) — temporary worsening of long standing ptsd from Vietnam experience
rise in PSA (Reproductive system and breast disorders) | 1 (1) | 0 (0) — patient had history of prostate cancer
gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) — patient given Prilosec for this
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — arthritis pain, periodic

LIMITATIONS AND CAVEATS:
The enrollment was very small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No